CLINICAL TRIAL: NCT04589910
Title: What Are Reference Values of the Thickness and the Thickening Fraction of the Diaphragm in Children Aged 0-8 Years?
Brief Title: Measuring Thickness of the Normal Diaphragm in Children Via Ultrasound.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Erasmus Medical Center (Other)
Responsible Party: Principal Investigator, Erwin Ista, PhD, Associate professor nursing science, Erasmus Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: NL70476.078.19
Record Dates: First submitted 2020-10-09; First posted 2020-10-19 (Actual); Last update posted 2022-08-12 (Actual); Status verified 2022-08

CONDITIONS: Mechanical Ventilation Complication; Pediatric ALL; Intensive Care Unit Acquired Weakness
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Ultra-sound arm (Other): Ultrasound measurement of the diaphragm will be performed with the use of a Sono Site SII, portable system in B mode with the child in a 30-degree supine position. The diaphragm thickness will be measured with a high frequency (4-10 MHz) linear array transducer placed in the ninth or tenth intercostal space between the anterior and midaxillary lines in the zone of apposition between lung and liver.
  Interventions: Diagnostic Test: diaphragm thickness and thickening fraction

INTERVENTIONS:
Diagnostic Test: diaphragm thickness and thickening fraction — Ultrasound measurement of the diaphragm will be performed with the use of a Sono Site SII, portable system in B mode with the child in a 30-degree supine position. The diaphragm thickness will be measured with a high frequency (4-10 MHz) linear array transducer placed in the ninth or tenth intercostal space between the anterior and midaxillary lines in the zone of apposition between lung and liver.

SUMMARY:
Critically ill children treated with invasive mechanical ventilation (iMV) in a paediatric intensive care unit (PICU) may suffer from complications leading to prolonged duration of ventilation and PICU stay. Prolonged ventilation is associated with haemodynamic dysfunction, neuromuscular insufficiency, malnutrition, metabolic disorders and diaphragmatic muscle weakness. Evidence from adult critical care supports the existence of ventilator induced diaphragmatic dysfunction, defined as a iMV-induced loss of diaphragmatic force - generating capacity - characterised by muscle fibre atrophy, myofibril necrosis and disorganization.

Diaphragm function or contractility can be assessed by measuring the diaphragm thickening during inspiration and expiration with ultrasound and is expressed as a thickening fraction (TF).

A low diaphragm contractile activity in adults has been associated with rapid decreases in diaphragm thickness, whereas high contractile activity has been associated with increases in diaphragm thickness. Contractile activity decreased with increasing ventilator driving pressure and controlled ventilator mode. Maximal thickening fraction (a measure of diaphragm function) was lower in patients with decreased as well as increased diaphragm thickness than in patients with unchanged thickness (p=0.05). Titrating ventilatory support to maintain normal levels of inspiratory effort may prevent changes in diaphragm configuration associated with iMV, but more research is needed to confirm this supposition.

Only one study has shown the presence of diaphragm atrophy in critically ill children on iMV for acute respiratory failure. The diaphragm contractility, measured as thickening fraction, was strongly correlated with a spontaneous breathing fraction.

Norm data for diaphragmatic thickness and TF in children are only available for healthy neonates (n=15) and children (n=48) from 8 till 20 years of age.

The purpose of this study is to determine values of normal diaphragm thickness and TF in children aged 0-8 years by ultrasound. This age range reflects the largest patient group treated in the PICU.

Once these values are known, the clinical relevance of the measuring of the diaphragm thickness of ventilated children by ultrasound can be further studied.

Objective of the study:

Primary objective: To determine diaphragm thickness and thickening fraction in healthy children below or equal to 8 years of age.

Secondary objective: To determine the interrater reliability of operators performing the ultra-sound

Study design:

prospective, cohort study.

Study population:

Healthy children in four age groups: 0-6 months; 6 months-1 year; 2-4 years; and 5-8 years.

Participants will be recruited in two ways:

Group 1. Parents of children scheduled to undergo a daycare procedure will asked permission for their child to join the study. These children undergo a minor procedure and are assumed to have a normal diaphragm; therefore are considered 'healthy''.

Group 2. Health professionals working on the PICU or other departments of Erasmus MC-Sophia as well as family, friends and neighbours of members of the research group will be asked to recruit 'healthy' children. The investigators will recruit participants by means of brochures in which children and/or caregivers are invited to contact the researchers when interested to participate in this study.

Primary study parameters/outcome of the study:

To determine diaphragm thickness and thickening fraction in healthy children below or equal to 8 years of age.

Secondary study parameters/outcome of the study (if applicable):

To determine the interrater reliability of operators performing the ultra-sound

ELIGIBILITY:
Inclusion Criteria:

Group 1

* Children aged 0-8 years old undergoing one of the following daycare procedures:
* Surgery: inguinal hernia and umbilical hernia surgery
* Urology: hypospadias surgery
* Throat/nose/ear surgery: tympanostomy tubes, removal of throat and nasal tonsils
* Orthopedics: congenital club feet surgery, hip luxation surgery, removing pins
* Plastic surgery: protruding ears surgery, removing of accessory auricle, removing additional toes and fingers - Ophthalmology: cataract and strabismus surgery
* Immunology: infusion therapy: e.g. prophylaxis of immunoglobulins

Group 2

-Children aged 0-8 years old recruited by colleagues, or relatives, friends and neighbours of members of the research group

Exclusion Criteria:

Neuromuscular diseases

* Lung diseases
* Recent abdominal or thoracic surgery (less than 3 month ago) - Deviations of the diaphragm

Ages: 0 Months to 8 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 120 (Actual)
Dates: Start 2020-09-01 (Actual); Primary Completion 2021-05-01 (Actual); Study Completion 2021-08-01 (Actual)

PRIMARY OUTCOMES:
diaphragm thickness | Day 1
  To determine diaphragm thickness and thickening fraction in healthy children below or equal to 8 years of age.

SECONDARY OUTCOMES:
Interrater reliability | During 6 months
  Interrater reliability of operators performing the ultra-sound

CONTACTS AND LOCATIONS:
Locations (1):
- Erasmus MC-Sophia Children's Hospital, Rotterdam, Netherlands

REFERENCES:
- [Derived] Duyndam A, Smit J, Heunks L, Molinger J, IJland M, van Rosmalen J, van Dijk M, Tibboel D, Ista E. Reference values of diaphragmatic dimensions in healthy children aged 0-8 years. Eur J Pediatr. 2023 Jun;182(6):2577-2589. doi: 10.1007/s00431-023-04920-6. Epub 2023 Mar 20. PMID 36939879